CLINICAL TRIAL: NCT03289351
Title: Randomized Control Trial: Two Different Antibiotics Versus One Antibiotic for Pediatric Perforated Appendicitis
Brief Title: Two Different Antibiotics Versus One Antibiotic for Pediatric Perforated Appendicitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-011
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-03

CONDITIONS: Perforated Appendicitis; Postoperative Infection
MeSH Terms: conditions — Appendicitis | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2-drug Therapy (No Intervention): ceftriaxone/metronidazole
- 1-drug Therapy (Experimental): piperacillin-tazobactam
  Interventions: Drug: Piperacillin, Tazobactam Drug Combination

INTERVENTIONS:
Drug: Piperacillin, Tazobactam Drug Combination — Single drug therapy
  Other Names: piperacillin-tazobactam; Zosyn
  Arms: 1-drug Therapy

SUMMARY:
After appendix has been removed for perforated appendicitis, patients will receive postoperative antibiotics. In the last 5 years, the literature has transitioned from a 3 -drug therapy to 2-drug therapy. Now there is a recent literature suggesting a single-drug therapy may be safe and adequate. In fact, using zosyn (piperacillin-tazobactam) as a single-drug therapy, there are additional benefits of simplicity, compliance, and lower infectious complications. Currently surgeons are already using both 2-drug regimen (ceftriaxone/metronidazole) and single-drug regimen (zosyn) interchangeable as both are FDA approved and regulated antibiotics for intra-abdominal infection. There is a clear need to compare outcomes between these two options.

DETAILED DESCRIPTION:
The diagnosis of perforated appendicitis will be documented intraoperatively with photos of extraluminal fecal contents or visible holes on the appendix. Patients will be randomized to 121 in each arm. Postoperative antibiotic therapy option will be decided based on blinded sequence model. 30 day postoperative follow up visit or calls will be made to assess and collect infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative Perforated Appendicitis (documented by intraoperative photo)
* Postoperative Laparoscopic Appendectomy

Exclusion Criteria:

* Nonperforated Gangrenous Appendicitis
* Nonperforated Purulent Appendicitis
* Open Appendectomy

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lee, MD, Principal Investigator — Phoenix Childrens Hospital
Locations (2):
- United States (2):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 2-drug Therapy: ceftriaxone/metronidazole - 2-drug regimen (CM) includes once a day dosing of ceftriaxone (50 mg/kg) and metronidazole (30 mg/kg)
- 1-drug Therapy: piperacillin-tazobactam - Single drug regimen (P) includes piperacillin-tazobactam (<40 kg: 100 mg/kg Q8HR, >40 kg: 3000mg Q6HR)
Period: Overall Study
Arm/Group | 2-drug Therapy | 1-drug Therapy
Started | 80 | 82
Completed | 80 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-drug Therapy | 1-drug Therapy | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 82 | 162
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 50 | 46 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 80 | 82 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Postoperative Intra-abdominal Abscess
Description: Intra-abdominal abscess documented by ultrasound or computerized tomography
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2-drug Therapy | 1-drug Therapy
Number analyzed (Participants) | 80 | 82
Participants | 19 | 5

2. Secondary Outcome: Number of Participants With Postoperative Surgical Site Infection
Description: surgical site infections including superficial port site infection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2-drug Therapy | 1-drug Therapy
Number analyzed (Participants) | 80 | 82
Participants | 4 | 4

3. Secondary Outcome: Number of Participants With a Postoperative Readmission
Description: readmission within 30 days for any gastrointestinal complaints or infectious complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 2-drug Therapy | 1-drug Therapy
Number analyzed (Participants) | 80 | 82
Participants | 11 | 4

ADVERSE EVENTS:
Time Frame: Assessed up to 30 days postoperatively.
Arm/Group | 2-drug Therapy | 1-drug Therapy
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/82
Other Adverse Events (participants affected / at risk) | 1/80 | 0/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-drug Therapy (N=80) | 1-drug Therapy (N=82)
Perioperative Redness/Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject developed perioperative redness and edema after operation. Originally given Zosyn which was discontinued and later replaced by another set of antibiotics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT03289351/Prot_SAP_000.pdf